CLINICAL TRIAL: NCT06958211
Title: A Phase 3, Double-Blind, Randomized, Vehicle-Controlled, Efficacy and Safety Study of Ruxolitinib Cream in Participants With Hidradenitis Suppurativa
Brief Title: Study to Evaluate the Efficacy and Safety of Ruxolitinib Cream in Participants With Hidradenitis Suppurativa (TRuE-HS2)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INCB018424-325; 2024-517633-40-00 (Registry Identifier: EU CT Number)
Record Dates: First submitted 2025-04-25; First posted 2025-05-06 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Hidradenitis Suppurativa
Keywords: Hidradenitis suppurativa; skin disease; ruxolitinb cream
MeSH Terms: conditions — Hidradenitis Suppurativa; Skin Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ruxolitinib 1.5 % Cream (Experimental): Participants received ruxolitinib 1.5% cream, applied topically to the affected area as defined in the protocol.
  Interventions: Drug: Ruxolitinib Cream
- Vehicle Cream (Placebo Comparator): Participants received vehicle cream, applied topically to the affected area as defined by the protocol.
  Interventions: Drug: Vehicle Cream

INTERVENTIONS:
Drug: Ruxolitinib Cream — Ruxolitinib cream applied topically to the affected area as a thin film twice daily.
  Arms: Ruxolitinib 1.5 % Cream
Drug: Vehicle Cream — Matching vehicle cream applied topically to the affected area as a thin film twice daily.
  Arms: Vehicle Cream

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of ruxolitinib cream in participants with hidradenitis suppurativa.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of HS for at least 6 months prior to screening visit.
* Mild to moderate HS (Hurley I or II) with the following at both screening and baseline visits:

  * A total AN count of at least 4, with no draining tunnels AND
  * Affecting at least 2 distinct anatomical areas
* Agreement to NOT use topical and systemic antibiotics for treatment of HS during the vehicle-controlled period.
* Agreement to NOT use topical antiseptics, including washes and leave-on products on the areas affected by HS lesions during the vehicle-controlled period and Weeks 16 to 20 of the extension period.
* Further inclusion criteria apply.

Exclusion Criteria:

* Body surface areas to be treated exceed 20% BSA at screening or baseline
* Presence of draining tunnels at screening or baseline.
* Medical history including current or history of certain infections, cancer, lymphoproliferative disorders and other medical conditions at the discretion of the investigator.
* Laboratory values outside of the protocol-defined criteria.
* Pregnant or lactating participants, or those considering pregnancy during the period of their study participation.
* Further exclusion criteria apply.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2025-06-12 (Actual); Primary Completion 2026-10-09 (Estimated); Study Completion 2027-07-11 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants who achieve Hidradenitis Suppurativa (HS) Clinical Response 75 (HiSCR75) from baseline | Week 16
  HiSCR75 is defined as at least a 75% reduction from baseline in the total abscess and/or inflammatory nodule (AN) count with no increase from baseline in abscess or draining tunnel count.

SECONDARY OUTCOMES:
Proportion of participants with ≥ 1 flare | Up to 16 weeks
  Defined as ≥ 25% increase in AN count with a minimum increase in total AN count of 2 relative to baseline.
Proportion of participants who achieve Skin Pain Numeric Rating Scale (NRS)30 among participants with baseline Skin Pain NRS score ≥ 3 | Week 16
  Participants with a Skin Pain score of at least 3 at baseline and who achieve Skin Pain NRS30, defined as at least a 30% reduction and at least 1-unit reduction from baseline in the Skin Pain NRS.
Treatment-IR Population: Proportion of participants who achieve Hidradenitis Suppurativa Clinical Response 75 (HiSCR75) from baseline | Week 16
  Treatment IR-Population defined as participants who had an inadequate response, intolerance, or contraindication to prior topical or systemic medications for HS. HiSCR75 is defined as at least a 75% reduction from baseline in the total AN count with no increase from baseline in abscess or draining tunnel count.
Treatment-IR Population: Proportion of participants with ≥ 1 HS flare | Up to 16 weeks
  Defined as ≥ 25% increase in total AN count with a minimum increase in AN count of 2 relative to baseline.
Treatment-IR Population: Proportion of participants who achieve Skin Pain Numeric Rating Scale (NRS)30 at Week 12 among participants with baseline Skin Pain NRS score ≥ 3 | Week 16
  Participants with a Skin Pain score of at least 3 at baseline and who achieve Skin Pain NRS30, defined as at least a 30% reduction and at least 1-unit reduction from baseline in the Skin Pain NRS.
Proportion of participants who achieve HiSCR50/75/90/100 at each postbaseline visit | Up to 16 weeks
  Defined as ≥ 50%/75%/90%/100% reduction from baseline in total AN count with no increase from baseline in abscess or draining tunnel count.
Extension Period: Proportion of participants with ≥ 1 HS flare | From Week 16 through Week 52
  Defined as ≥ 25% increase in total AN count with a minimum increase in AN count of 2 relative to baseline.
Proportion of participants who achieve abscess and/or inflammatory nodule (AN)75 at each postbaseline visit | Up to 52 weeks
  Defined as ≥ 75% reduction from baseline in total AN count.
Mean change from baseline in total AN count at each postbaseline visit | Up to 52 weeks
  Defined as mean change in total AN count.
Percentage change from baseline in total AN count at each postbaseline visit | Up to 52 weeks
  Defined as percent change from baseline in total AN count.
Mean change from baseline in abscess count at each postbaseline visit | Up to 52 weeks
  Defined as mean change of abscess(es) count relative to baseline.
Percentage change from baseline in abscess count at each postbaseline visit | Up to 52 weeks
  Percent Change from baseline in number of abscess(es).
Mean change from baseline in inflammatory nodule count at each postbaseline visit | Up to 52 weeks
  Defined as mean change of inflammatory nodule count relative to baseline.
Percentage change from baseline in inflammatory nodule count at each postbaseline visit | Up to 52 weeks
  Defined as percent change from baseline in number of inflammatory nodule(s).
Proportion of participants with presence of draining tunnels at each postbaseline visit | Up to 52 weeks
  Participants with presence of draining tunnels.
Proportion of participants who achieve Skin Pain Numeric Rating Scale (NRS)30 among participants with baseline Skin Pain NRS score ≥ 3 at each postbaseline visit | Up to 52 weeks
  Participants with a Skin Pain score of at least 3 at baseline and who achieve Skin Pain NRS30, defined as at least a 30% reduction and at least 1-unit reduction from baseline in the Skin Pain NRS.
Proportion of participants who achieve Itch Numeric Rating Scale (NRS)30 among participants with baseline Itch NRS score ≥ 3 at each postbaseline visit | Up to 52 weeks
  Participants with a Itch score of at least 3 at baseline and who achieve Itch NRS30, defined as at least a 30% reduction and at least 1-unit reduction from baseline in the Itch NRS.
Proportion of participants who achieve Patient Global Impression of Change (PGIC) at each postbaseline visit | Up to 52 weeks
  The PGIC is based on a 7-point scale and the participant will rate each question from the start of treatment as 1-very much improved, 2-much improved, 3-minimally improved, 4-no change, 5-minimally worse, 6-much worse, and 7-very much worse.
Proportion of participants who achieve PGIC score 1 or 2 at each postbaseline visit | Up to 52 weeks
  The PGIC is based on a 7-point scale and the participant will rate each question from the start of treatment as 1-very much improved, 2-much improved, 3-minimally improved, 4-no change, 5-minimally worse, 6-much worse, and 7-very much worse.
Patient Global Impression of Severity (PGIS) score at each postbaseline visit | Up to 52 weeks
  The PGIS is a single-item, self-reporting measure in which the participant rates the severity of their overall status over the past week based on a 5-point scale: (1) none, (2) mild, (3) moderate, (4) severe, and (5) very severe.
Change from baseline in PGIS Score at each postbaseline visit | Up to 52 weeks
  The PGIS is a single-item, self-reporting measure in which the participant rates the severity of their overall status over the past week based on 5-point scale: (1) none, (2) mild, (3) moderate, (4) severe, and (5) very severe.
Proportion of participants who achieve status of Dermatology Life Quality Index (DLQ1)4 at each postbaseline visit | Up to 52 weeks
  Defined as a ≥ 4-point reduction in DLQI score relative to baseline. The DLQI is a simple, 10-question, validated questionnaire to measure how much a skin problem has affected an adult participant over the previous 7 days, across symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment.
Proportion of participants who achieve status of Children's Dermatology Life Quality Index (CDLQ1)6 at each postbaseline visit | Up to 52 weeks
  Defined as a ≥ 6-point reduction in CDLQI score relative to baseline. The CDLQI is a 10-question, validated questionnaire to measure the impact of skin disease on the lives of children over the previous 7 days.
Change from baseline in Hidradenitis Suppurativa Quality of Life (HiSQoL) score at each postbaseline visit | Up to 52 weeks
  The HiSQoL is a 17-item, HS-specific, health-related, quality-of-life instrument with a 7-day recall period used to assess HS symptoms and the impact of HS problems on quality of life.
Percent change from baseline in Hidradenitis Suppurativa Quality of Life (HiSQoL) score at each postbaseline visit | Up to 52 weeks
  The HiSQoL is a 17-item, HS-specific, health-related, quality-of-life instrument with a 7-day recall period used to assess HS symptoms and the impact of HS problems on quality of life.
Change from baseline in Hidradenitis Suppurativa Quality of Life - Adolescent (HiSQoL-AA) at each postbaseline visit | Up to 52 weeks
  The HiSQoL-AA is a 15-item instrument with a 7-day recall period used to assess HS symptoms and experiences of HS in adolescent.
Percent change from baseline in Hidradenitis Suppurativa Quality of Life - Adolescent (HiSQoL-AA) at each postbaseline visit | Up to 52 weeks
  The HiSQoL-AA is a 15-item instrument with a 7-day recall period used to assess HS symptoms and experiences of HS in adolescent.
Change from baseline in EuroQol 5-dimension 5-level scale (EQ-5D-5L) score at each postbaseline visit | Up to 52 weeks
  The EQ-5D-5L questionnaire is a standardized, validated instrument for use as a measure of health outcome.
Treatment-IR Population: Change from baseline in total abscess count at each postbaseline visit | Up to 52 weeks
  Defined as change from baseline in total abscess count.
Treatment-IR Population: Percent change from baseline in total abscess count at each postbaseline visit | Up to 52 weeks
  Percent Change from baseline in total abscess count.
Treatment-IR Population: Change from baseline in total inflammatory nodule count at each postbaseline visit | Up to 52 weeks
  Defined as change from baseline in total number of inflammatory nodule(s).
Treatment-IR Population: Percent change from baseline in total inflammatory nodule count at each postbaseline visit | Up to 52 weeks
  Defined as percent change from baseline in number of inflammatory nodule(s).
Treatment-IR Population: Proportion of participants with presence of draining tunnels at each postbaseline visit | Up to 52 weeks
  Participants with presence of draining tunnels.
Number of Treatment Emergent Adverse Events (TEAEs) | Up to 56 weeks
  A TEAE or treatment emergent SAE is any AE or SAE either reported for first time or worsening of a pre-existing event after first application of study cream.

CONTACTS AND LOCATIONS:
Overall Officials: Incyte Study Monitor, Study Director — Incyte Corporation
Locations (110):
- United States (70):
  - Investigative Site US257, Birmingham, Alabama
  - Investigative Site US218, Birmingham, Alabama
  - Investigative Site US239, Montgomery, Alabama
  - Investigative Site US215, Phoenix, Arizona
  - Investigative Site US261, Phoenix, Arizona
  - Investigative Site US221, Scottsdale, Arizona
  - Investigative Site US240, Tucson, Arizona
  - Investigative Site US262, Encino, California
  - Investigative Site US222, Fountain Valley, California
  - Investigative Site US211, Los Angeles, California
  - Investigative Site US237, Los Angeles, California
  - Investigative Site US234, Northridge, California
  - Investigative Site US250, Santa Ana, California
  - Investigative Site US244, Castle Rock, Colorado
  - Investigative Site US252, Cromwell, Connecticut
  - Investigative Site US208, Boca Raton, Florida
  - Investigative Site US203, Hialeah, Florida
  - Investigative Site US258, Jacksonville, Florida
  - Investigative Site US206, Maitland, Florida
  - Investigative Site US223, Miami, Florida
  - Investigative Site US241, Miami, Florida
  - Investigative Site US202, Miami, Florida
  - Investigative Site US214, Tampa, Florida
  - Investigative Site US247, Tampa, Florida
  - Investigative Site US231, Columbus, Georgia
  - Investigative Site US225, Sandy Springs, Georgia
  - Investigative Site US233, Ketchum, Idaho
  - Investigative Site US207, Skokie, Illinois
  - Investigative Site US205, Plainfield, Indiana
  - Investigative Site US264, Lake Charles, Louisiana
  - Investigative Site US326, New Orleans, Louisiana
  - Investigative Site US266, New Orleans, Louisiana
  - Investigative Site US254, Gambrills, Maryland
  - Investigative Site US201, Marriottsville, Maryland
  - Investigative Site US253, Milford, Massachusetts
  - Investigative Site US227, Needham, Massachusetts
  - Investigative Site US268, Worcester, Massachusetts
  - Investigative Site US238, Ann Arbor, Michigan
  - Investigative Site US230, Auburn Hills, Michigan
  - Investigative Site US251, St Louis, Missouri
  - Investigative Site US271, Wildwood, Missouri
  - Investigative Site US212, Missoula, Montana
  - Investigative Site US216, Las Vegas, Nevada
  - Investigative Site US235, Hoboken, New Jersey
  - Investigative Site US217, Albuquerque, New Mexico
  - Investigative Site US219, Brooklyn, New York
  - Investigative Site US246, Elmhurst, New York
  - Investigative Site US269, Fairport, New York
  - Investigative Site US213, Kew Gardens, New York
  - Investigative Site US242, New York, New York
  - Investigative Site US245, Rochester, New York
  - Investigative Site US259, Huntersville, North Carolina
  - Investigative Site US263, Winston-Salem, North Carolina
  - Investigative Site US228, Cleveland, Ohio
  - Investigative Site US243, Columbus, Ohio
  - Investigative Site US249, Columbus, Ohio
  - Investigative Site US204, Portland, Oregon
  - Investigative Site US226, Plymouth Meeting, Pennsylvania
  - Investigative Site US256, Bluffton, South Carolina
  - Investigative Site US267, Mt. Pleasant, South Carolina
  - Investigative Site US255, Austin, Texas
  - Investigative Site US260, Cypress, Texas
  - Investigative Site US270, Prosper, Texas
  - Investigative Site US232, Sugar Land, Texas
  - Investigative Site US248, Arlington, Virginia
  - Investigative Site US209, Danville, Virginia
  - Investigative Site US229, Norfolk, Virginia
  - Investigative Site US265, Seattle, Washington
  - Investigative Site US224, Spokane, Washington
  - Investigative Site US210, Milwaukee, Wisconsin
- Belgium (4):
  - Investigative Site BE204, Brussels
  - Investigative Site BE201, Ghent
  - Investigative Site BE203, Ghent
  - Investigative Site BE202, Leuven
- Bulgaria (3):
  - Investigative Site BG201, Sevlievo
  - Investigative Site BG202, Sofia
  - Investigative Site BG203, Sofia
- Canada (9):
  - Investigative Site CA209, Edmonton, Alberta
  - Investigative Site CA201, Winnipeg, Manitoba
  - Investigative Site CA207, Fredericton, New Brunswick
  - Investigative Site CA202, Hamilton, Ontario
  - Investigative Site CA203, London, Ontario
  - Investigative Site CA204, Markham, Ontario
  - Investigative Site CA205, Mississauga, Ontario
  - Investigative Site CA208, Saskatoon, Saskatchewan
  - Investigative Site CA206, St. John's
- France (4):
  - Investigative Site FR201, Reims
  - Investigative Site FR203, Rouen
  - Investigative Site FR204, Saint-Etienne
  - Investigative Site FR202, Toulouse
- Germany (6):
  - Investigative Site DE207, Bad Bentheim
  - Investigative Site DE206, Göttingen
  - Investigative Site DE202, Hanover
  - Investigative Site DE203, Kiel
  - Investigative Site DE205, Langenau
  - Investigative Site DE204, Merzig
- Netherlands (2):
  - Investigative Site NL203, Amsterdam
  - Investigative Site NL201, Rotterdam
- Poland (4):
  - Investigative Site PL202, Lublin
  - Investigative Site LP204, Poznan
  - Investigative Site PL201, Rzeszów
  - Investigative Site PL203, Wroclaw
- Spain (8):
  - Investigative Site ES205, Barcelona
  - Investigative Site ES208, Esplugues de Llobregat
  - Investigative Site ES201, Granada
  - Investigative Site ES206, Granollers
  - Investigative Site ES202, Las Palmas de Gran Canaria
  - Investigative Site ES203, Madrid
  - Investigative Site ES207, Manises
  - Investigative Site ES204, Santiago de Compostela

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency

REFERENCES:
- See also: Study to Evaluate the Efficacy and Safety of Ruxolitinib Cream in Participants With Hidradenitis Suppurativa (TRuE-HS2) — https://incyteclinicaltrials.com/studies/incb018424-325